CLINICAL TRIAL: NCT06130774
Title: Effects of Retro-walking in Knee OA Along With Conventional Therapy
Brief Title: Effects of Retro-walking in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01681 MAIRA KANWAL
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Osteo Arthritis Knee
Keywords: osteoarthritis; retrowalking; balance; gait
MeSH Terms: conditions — Osteoarthritis | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retro walking and conventional (Experimental): Patient will start retro walking with first he/she will raise his/her one foot with toe off first then heel will be off from ground. swing phase of same leg would be done in backward direction with flexion on knee and extension will be performed on hip. Then patient will place the same foot on ground behind the other foot, with toe touch first on ground, and so this way patient would continue for 20 minutes continue his retro-walk for 20 minutes.
  Interventions: Other: Retro walking and conventional
- conventional therapy (Active Comparator): Hot pack in supine lying (10min) TENS (10min ) Tibiofemoral mobilization (grade 1,2 ,3) (10rep) Static quadriceps exercise in supine (10rep x 3sec x2set) hip abduction in side lying(10repx 2set) knee bending exercise in prone lying ( 10rep x 2set) Hamstring stretch in supine ( 10 rep x 2 set)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Retro walking and conventional — Patient will start retro walking with first he/she will raise his/her one foot with toe off first then heel will be off from ground. swing phase of same leg would be done in backward direction with flexion on knee and extension will be performed on hip. Then patient will place the same foot on ground behind the other foot, with toe touch first on ground, and so this way patient would continue his retro-walk for 20 minutes
  Arms: Retro walking and conventional
Other: conventional therapy — Hot pack in supine lying (10min) TENS (10min ) Tibiofemoral mobilization (grade 1,2 ,3) (10rep) Static quadriceps exercise in supine (10rep x 3sec x2set) hip abduction in side lying(10repx 2set) knee bending exercise in prone lying ( 10rep x 2set) Hamstring stretch in supine ( 10 rep x 2 set)
  Arms: conventional therapy

SUMMARY:
Osteoarthritis is degenerative joint disease that cause deterioration of the articular cartilage and neighboring tissue and lead to osteophyte formation, weakening of surrounding muscles, ligamentous laxity and inflammation of synovium. Diagnosis can be made based on history and clinical features and risk factors including age, sex, body mass index , absence of whole leg pain, fixed flexion deformity, absence of traumatic event, restricted flexion range of motion, pain in descending stairs, palpable effusion and crepitus. Confirmation is usually based on radiological finding according to Kellgren and Lawrence diagnostic scale . Radio graphic changes of osteoarthritis of the knee are bilateral in 85% of patients .

DETAILED DESCRIPTION:
Knee pain is a major symptom of knee osteoarthritis (OA) that lead to stiffness, and capsular contracture along with muscle spasm. Decreased flexibility of muscles reduces the joint range of motion and thus contributes to increase in the stiffness of the joint lead to physical disability in persons with knee OA.Eighty percent of persons with knee OA experience pain and 25% struggle to perform activities of daily living.) Retro-walking is sometimes referred to as backward walking, has been thought to be used already for several decades in China, Japan and Europe to get a physical workout, improve sport performance, promote balance and also to stay mentally fit .

In fact in Europe, they have races which vary from sprints to the 26.2 miles marathon.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Knee OA .
* Kellgren-Lawrence grading (grade 1 and 2)
* Participants fulfilling three out of the six clinical criteria listed by the American College of Rheumatology The criteria are Age >40 years, Morning stiffness lasting <30 mins. Crepitus with active motion, Bony tenderness, Bony enlargement and No warmth to touch and diagnosed to have knee OA
* Pain more than 6 weeks

Exclusion Criteria:

* Trauma or surgery in the last 6 months.
* Hip, knee, and foot deformities.
* Stroke and other neurovascular issues.
* Severe pain (greater than 7 in NPRS)
* Difficulty in walking for 10 min continuously.
* Obesity (body mass index greater than 25 kg/m2 )
* Osteoporosis
* Patients having any systemic joint pathology, inflammatory joint disease (e.g. rheumatoid arthritis, gouty arthritis, psoriatic arthritis).
* Patients who had any neurological deficit, myelopathy any mental illness.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
NPRS | six weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. NPRS exhibited moderate reliability
WOMAC | six weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68),
Calcon Calculator | six weeks
  To calculate your walking stride length, divide the number of steps you took by two and divide that number into the measured distance. If it took you 18 steps to cover 21 feet, divide the number of steps (18) by 2 to get the number of strides. Then take the answer (9) and divide it into the distance. Distance in feet/number of strides = stride length. In this case, you took nine strides in 22 feet, so your stride length would be 2.4 feet. For step length divide the number of steps into the measured distance. Distance in feet/number of steps = step length.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international hospital Sihala, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No